CLINICAL TRIAL: NCT03957057
Title: Randomized Trial Comparing Intravenous Iron Carboxymaltose, Intravenous Iron Isomaltoside and Oral Iron Sulphate for Postpartum Anemia
Brief Title: Intravenous Iron Carboxymaltose, Isomaltoside and Oral Iron Sulphate for Postpartum Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Miha Lucovnik, assistant professor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-117/2019/5
Record Dates: First submitted 2019-05-14; First posted 2019-05-21 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Postpartum Anemia Nos; Iron-deficiency
Keywords: postpartum anemia; iron deficiency; ferrous sulphate; ferric carboxymaltose; ferric isomaltoside
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — ferric carboxymaltose; iron isomaltoside 1000; ferrous sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Iron carboxymaltose group (Experimental): Iron carboxymaltose group. Total dose of intravenous ferric carboxymaltose (Iroprem®) needed to correct anemia and replenish iron stores will be calculated using the Ganzoni formula (28) modified to include adjustment for baseline iron status: prepregnancy weight in kilograms X (15-baseline Hb) X 2.4 + 500. Fifteen is the target Hb in g/dL, 2.4 is a unit less conversion constant and 500 is the target iron stores in mg. The maximal dose administered in a single day will not exceed 15 mg/kg (current weight) or 1000 mg (for participants with body weight > 67 kg). If total calculated dose will exceed 15 mg/kg or 1000 mg, subsequent doses will be administered weekly until the total calculated dose will be reached.
  Interventions: Drug: Iron Carboxymaltose
- Iron isomaltoside group (Experimental): Total dose of intravenous iron isomaltoside (Monofer®) needed to correct anemia and replenish iron stores will be calculated as described above. The maximal dose administered in a single day will not exceed 20 mg/kg (current weight) or 1500 mg (for participants with body weight > 75 kg). If total calculated dose will exceed 20 mg/kg or 1500 mg, subsequent doses will be administered weekly until the total calculated dose will be reached.
  Interventions: Drug: Iron Isomaltoside
- Iron sulphate group (Active Comparator): Iron sulphate group. Participants will receive oral ferrous sulphate (Tardyfer®) 160 mg daily for 6 weeks with instruction to take two tablets by mouth once daily 1 hour before meal. They will receive no additional iron supplementation.
  Interventions: Drug: Ferrous sulphate

INTERVENTIONS:
Drug: Iron Carboxymaltose — Intravenous iron carboxymaltose application
  Arms: Iron carboxymaltose group
Drug: Iron Isomaltoside — Inravenous iron isomaltoside application
  Arms: Iron isomaltoside group
Drug: Ferrous sulphate — Oral ferrous sulphate application
  Arms: Iron sulphate group

SUMMARY:
Anemia affects between 20 and 50 % of women in the postpartum period. It is associated with several adverse health consequences, such as impaired physical work capacity, deficits in cognitive function and mood, reduced immune function and reduced duration of breastfeeding. Postpartum anemia has also been shown to be a major risk factor for postpartum depression and to significantly disrupt maternal-infant interactions. Iron deficiency is the principal cause of anemia after delivery. Oral iron supplementation with ferrous sulfate has been considered the standard of care with blood transfusion reserved for more severe or symptomatic cases. In the last decade, two new intravenous iron compounds have been registered for clinical use: ferric carboxymaltose (Iroprem®) and iron isomaltoside (Monofer®). No study to date compared efficacy of iron carboxymaltose to iron isomaltoside for treatment of postpartum anemia.

The objective of the study is to compare efficacy of intravenous iron carboxymaltose to intravenous iron isomaltoside and oral iron sulphate for treatment of postpartum anemia.

DETAILED DESCRIPTION:
RATIONALE Anemia affects between 20 and 50 % of women in the postpartum period. It is associated with several adverse health consequences, such as impaired physical work capacity, deficits in cognitive function and mood, reduced immune function and reduced duration of breastfeeding. Postpartum anemia has also been shown to be a major risk factor for postpartum depression and to significantly disrupt maternal-infant interactions.

Iron deficiency is the principal cause of anemia after delivery. Oral iron supplementation with ferrous sulfate has been considered the standard of care with blood transfusion reserved for more severe or symptomatic cases. However, efficacy of oral iron is limited by gastrointestinal side effects, patient non-adherence as well as prolonged time required to treat anemia and replenish body iron stores. Blood transfusion, on the other hand, is associated with several hazards, including transfusion of the wrong blood type, infection, anaphylaxis and lung injury.

In last decades, modern formulations of intravenous iron have emerged as safe and effective alternatives to oral iron supplementation for iron deficiency anemia management outside pregnancy. Several studies have also evaluated efficacy of intravenous iron preparations for treatment of postpartum anemia. Westad et al. reported no significant difference in hemoglobin levels at 4, 8 and 12 weeks postpartum in women receiving intravenous iron sucrose (Venofer®) compared to those receiving oral ferrous sulphate, whereas the total fatigue score was significantly improved in the intravenous iron supplementation group at weeks 4, 8 and 12. In addition, mean serum ferritin value after 4 weeks was significantly higher in the iron sucrose group. Several other authors came to similar conclusion, intravenous iron sucrose and oral ferrous sulphate were both effective in correcting peripartum anemia, although intravenous iron restored stores faster than oral iron.

In the last decade, two new intravenous iron compounds have been registered for clinical use: ferric carboxymaltose (Iroprem®) and iron isomaltoside (Monofer®). These treatments were designed to be administered in large doses by rapid intravenous injection. They have been demonstrated to be more efficacious than intravenous iron sucrose in patients with inflammatory bowel disease and in patients with chronic kidney disease. In the postpartum period, ferric carboxymaltose has been compared to oral iron supplements in four randomized trials. All reported a faster rise in hemoglobin levels compared to oral ferrous sulphate. Pfenninger et al. compared efficacy of intravenous ferric carboxymaltose with iron sucrose for the treatment of postpartum anemia in a retrospective cohort study. Both drugs offered rapid normalization of hemoglobin levels after delivery with no difference in mean daily hemoglobin increase between the groups up to 8 days after treatment. Only one randomized study to date compared intravenous ferric carboxylase to intravenous iron sucrose and oral ferrous sulphate for treatment of postpartum anemia. Radhod et al. found a significantly faster rise in hemoglobin and ferritin levels with ferric carboxylase compared to iron sucrose and ferrous sulphate in Indian women presenting with anemia after delivery. This study, like most randomized trials on efficacy of various iron treatments, focused solely on hematological biomarkers. However, iron deficiency, even without anemia, contributes significantly to fatigue experienced by women in the puerperium, and these women may benefit from iron supplementation as well. Data on patient reported outcomes associated with different iron treatments are, therefore, very much needed. Holm et al. compared the effects of single-dose intravenous iron isomaltoside to oral iron supplementation on physical fatigue in women after postpartum haemorrhage. They found significant reduction in fatigue within 12 weeks postpartum in women who received iron isomaltoside. Iron isomaltoside treatment was also associated with improved haematological and iron parameters compared to oral ferrous sulfate.

No study to date, however, compared efficacy of iron carboxymaltose to iron isomaltoside for treatment of postpartum anemia. The only head-to-head comparison between these two compounds merely examined economic aspects of each treatment, showing potential reduction of costs associated with the use of iron isomaltoside vs. iron carboxymaltose.

OBJECTIVE The objective of the study is to compare efficacy of intravenous iron carboxymaltose to intravenous iron isomaltoside and oral iron sulphate for treatment of postpartum anemia.

METHODS Single-center, randomized, open-label trial.

After signed informed consent patients will be allocated randomly in a 1:1:1 fashion into one of three groups:

1. Iron carboxymaltose group. Total dose of intravenous ferric carboxymaltose (Iroprem®) needed to correct anemia and replenish iron stores will be calculated using the Ganzoni formula modified to include adjustment for baseline iron status: prepregnancy weight in kilograms X (15-baseline Hb) X 2.4 + 500. Fifteen is the target Hb in g/dL, 2.4 is a unit less conversion constant and 500 is the target iron stores in mg. The maximal dose administered in a single day will not exceed 15 mg/kg (current weight) or 1000 mg (for participants with body weight > 67 kg). If total calculated dose will exceed 15 mg/kg or 1000 mg, subsequent doses will be administered weekly until the total calculated dose will be reached.
2. Iron isomaltoside group. Total dose of intravenous iron isomaltoside (Monofer®) needed to correct anemia and replenish iron stores will be calculated as described above. The maximal dose administered in a single day will not exceed 20 mg/kg (current weight) or 1500 mg (for participants with body weight > 75 kg). If total calculated dose will exceed 20 mg/kg or 1500 mg, subsequent doses will be administered weekly until the total calculated dose will be reached.
3. Iron sulphate group. Participants will receive oral ferrous sulphate (Tardyfer®) 160 mg daily for 6 weeks with instruction to take two tablets by mouth once daily 1 hour before meal. They will receive no additional iron supplementation.

The investigators will monitor blood pressure and record adverse events in all patients before and after administration of IV iron and ask all patients to report any untoward medical event at its onset.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum patients with a hemoglobin level between 70 g/L and 100 g/L within 48 hours after delivery.

Exclusion Criteria:

* Contraindications for any of the study drugs.
* Anemia due to causes other than iron deficiency.
* Signs of systemic infection.
* Renal or hepatic dysfunction.
* Depression during pregnancy or pre-existing depressive disorders.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pospartum women will be included in the study.
Enrollment: 300 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Multidimensional Fatigue Inventory (MFI) score | 6 weeks postpartum
  Multidimensional Fatigue Inventory (MFI) score at 6 weeks postpartum. The MFI is a 20-item self-report instrument designed to measure fatigue. Items are scored 1-5, with 10 positively phrased items reverse scored (this concerns following items: 2, 5, 9, 10, 13, 14, 16, 17, 18, 19). For each of the 5 scales (general fatigue, physical fatigue, reduced activity, reduced motivation, and mental fatigue) a total score is calculated by summation of the scores of the individual items. Scores can range from the minimum of 4 to the maximum of 20. Higher scores indicate a higher degree of fatigue.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) score | 6 weeks postpartum
  Edinburgh Postnatal Depression Scale (EPDS) score at 6 weeks postpartum. EPDA is a 10-item questionnaire which evaluates different depression symptoms, such as guilt feeling, sleep disturbance, low energy, anhedonia, and suicidal ideation. Overall assessment is done by total score, which is determined by adding together the scores for each of the 10 items. Each answer is given a score of 0 to 3 . The maximum score is 30. Higher scores indicate more depressive symptoms. A score of more than 10 suggests minor or major depression may be present.
hemoglobin | 6 weeks postpartum
  Mean hemoglobin level at 6 weeks postpartum
hemoglobin level > 120 g/L | 6 weeks postpartum
  Proportion of participants with hemoglobin level > 120 g/L at 6 weeks postpartum
ferritin level > 50 mcg/L at 6 weeks postpartum | 6 weeks postpartum
  Proportion of participants with ferritin level > 50 mcg/L
reticulocyte count | 6 weeks postpartum
  Mean reticulocyte count
ferritin level | 6 weeks postpartum
  Mean ferritin level
transferrin level | 6 weeks postpartum
  Mean transferrin level
Costs of medication used in each study arm | 6 weeks postpartum
  Costs of treatments
Compliance - proportion of participants receiving treatments as recommended | 6 weeks postpartum
  Compliance with oral ferrous sulphate treatment
Side effects - proportion of participants reporting side effects of treatments | 6 weeks postpartum
  Side effects of all three study treatments in mothers (e.g. constipation, headache, infusion site burning) and infants (e.g. constipation, erythema, diarrhea, abdominal pain, upper respiratory tract infection)

CONTACTS AND LOCATIONS:
Overall Officials: Miha Lucovnik, MD, PhD, Principal Investigator — UMC Ljubljana
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will be willing to share IPD after study completion.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT03957057/Prot_SAP_000.pdf